CLINICAL TRIAL: NCT05276271
Title: The Effect of Levetiracetam Therapy on Lipid Profile in Epileptic Children
Brief Title: The Effect of Levetiracetam on Lipid Profile in Children
Status: Completed | Type: Observational
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, İpek Dokurel, Principal Investigator, Ege University
Other Study IDs: 2021/186
Record Dates: First submitted 2022-02-19; First posted 2022-03-11 (Actual); Last update posted 2022-03-11 (Actual); Status verified 2022-03

CONDITIONS: Epilepsy; Child, Only; Thyroid; Lipid Disorder
Keywords: Child; Epilepsy; Thyroid Hormones; Lipids
MeSH Terms: conditions — Epilepsy; Thyroid Diseases; Lipid Metabolism Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — The blood sample tests (TSH, fT3, fT4, TG, HDL, LDL, total cholesterol, AST, ALT, uric acid, CRP) for each enrolled patient and control subject were obtained the time after overnight fasting (at least 10 hours) at the outpatient clinic's admission.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- epileptic children: epileptic children who had been diagnosed with epilepsy with at least two focal seizures within a year, and treated with levetiracetam monotherapy for at least 12 months
  Interventions: Diagnostic Test: the blood sample test results
- healthy controls: healthy controls who was without an exposure to levetiracetam
  Interventions: Diagnostic Test: the blood sample test results

INTERVENTIONS:
Diagnostic Test: the blood sample test results — Retrospectively the fasting blood samples results were obtained for serum thyroid-stimulating hormone (TSH), free triiodothyronine, free thyroxine, total cholesterol (TC), high-density lipoprotein (HDL), low-density lipoprotein (LDL), triglycerides, Triglyceride/HDL Index, uric acid, CRP, and transaminases at the administration.
  Other Names: retrospectively collect the blood sample test results

SUMMARY:
Levetiracetam is a widely prescribed antiseizure medication in epileptic children due to an estimated better safety profile and easy accessibility. There is limited and contradicting data about the effect of levetiracetam on serum lipid metabolisms, especially in epileptic children. The aim of our study was to evaluate the effect of levetiracetam therapy on lipid metabolism in euthyroid non-obese epileptic children. In this case-control study, the investigators recruited 37 epileptic children receiving levetiracetam monotherapy for at least 12 months and 54 healthy controls. All the participants were euthyroid and within normal nutritional status limits for their age. Fasting blood samples were obtained for serum thyroid-stimulating hormone (TSH), free triiodothyronine, free thyroxine, total cholesterol (TC), high-density lipoprotein (HDL), low-density lipoprotein (LDL), triglycerides, Triglyceride/HDL Index, uric acid, CRP, and transaminases at the administration. The investigators would like to show if epileptic children with levetiracetam monotherapy are susceptible to lipid metabolism alterations.

DETAILED DESCRIPTION:
A total of 37 pediatric epileptic patients (children = 16, adolescents = 21) and 54 healthy control (children = 17, adolescents = 37) were enrolled to the study. Participants admitted to the pediatric neurology outpatient clinic of Ataturk City Hospital from October 2020 to October 2021 were recruited to this observational case-control study.

The pediatric neurologist and pediatric endocrinologist evaluated all the participants' medical data to determine their medical history and physical examination. Retrospectively, all the participants' age, gender, anthropometric assessments, BMI (body weight/height2), pubertal development staging, laboratory workup (thyroid-stimulating hormone (TSH), free triiodothyronine (fT3), free thyroxine (fT4), triglycerides (TG), high-density lipoprotein (HDL), low-density lipoprotein (LDL), total cholesterol (TC), aspartate aminotransferase (AST), alanine aminotransferase (ALT), uric acid, CRP) noted from the medical records. Height and weight measurements of the participants were made with a digital Harpenden stadiometer by the same person.

Seizure and epilepsy types of patients were categorized according to recommendations of the International League Against Epilepsy, 2017.

The degree of seizure control was categorized 'controlled' if they were seizure-free for ≥1 year, 'partially controlled' if the seizures' intervals were longer than seven days but shorter than 30 days, and 'uncontrolled' if the seizures occurred several times a day or at intervals shorter than seven days.

The Puberty Development Scale categorized in boys with testicular volume (testicular volume measured with a prader orchidometer) greater than 4 milliliters were considered pubertal. And for girls with breast development at Tanner stage 2 (breast development with an elevation of breast and papilla; enlargement of the areola) and above were considered pubertal.

All participants were established 'euthyroid' by evaluating TSH (mIU/L), fT3 (pmol/L), fT4(pmol/L). For participants aged 4-11.9 years, normal thyroid hormone levels were 0.2- 3.0 mIU/L for TSH, 4.6-8.2 pmol/L for fT3, and 13.8-35.3 pmol/L for fT4.For participants aged older than 11.9 years, published thyroid hormone values of Campbell et al. were used to determine normal thyroid hormone levels23. The physical examinations, blood tests (TSH, fT3, fT4, TG, HDL, LDL, total cholesterol, AST, ALT, uric acid, CRP) for each enrolled patient and control subject were obtained the time after overnight fasting (at least 10 hours) at the outpatient clinic's admission. Published lipid levels of the National Cholesterol Education Program guidelines were used for all participants 24. The TG/HDL index was calculated as the ratio of TG (mg/dL) to HDL (mg/dL) value.

The informed consent form was obtained from parents of all the children and healthy controls. The regional Ethics Committee approved the current study (2021/186-08/09/21). Statistical Analysis Statistical analyses were performed using the SPSS software version 25.0 (SPSS Statistics for Windows, 2017). The sample size was calculated by using the statistical software (G*Power version 3). The variables were investigated using visual (histogram, probability plots) and analytical methods (Kolmogorov-Smirnov) to determine whether they are normally distributed. Descriptive analyses were presented (using frequencies for ordinal variables) and using mean and standard deviation. Continuous variables were compared among the two groups by using an independent t-test. If the variable did not have a normal distribution, the Mann-Whitney U test was applied for the groups. A Chi-Square test was used to examine the association between categorical variables. A 5% type- I error level was used to infer statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Must be aged between 4 and 17 years
* Must be diagnosed with epilepsy with at least two focal seizures within a year
* Must be treated with levetiracetam monotherapy for at least 12 months.

Exclusion Criteria:

* other medical conditions requiring continuous medication
* abnormal thyroid function
* progressive neurologic conditions
* abnormal nutritional status (malnutrition, over-weight or obese)
* epilepsy requiring poly-therapy
* genetic diseases causing unbalanced laboratory and hormone profile

Ages: 1 Year to 18 Years | Sex: All
Age Groups: Child, Adult
Study Population: A total of 37 pediatric epileptic patients (children = 16, adolescents = 21) and 54 healthy control (children = 17, adolescents = 37) were enrolled to the study. Participants admitted to the pediatric neurology outpatient clinic of Ataturk City Hospital from October 2020 to October 2021 were recruited to this observational case-control study.
Sampling Method: Non-Probability Sample
Enrollment: 91 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-10-01 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
the effect of levetiracetam therapy on lipid profile | 1 year
  Lipid profile of the epileptic children who had been receiving levetiracetam monotherapy would be compared with the healthy controls

CONTACTS AND LOCATIONS:
Locations (1):
- Ataturk City Hospital, Altınoluk, Balikesi̇r, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
According to the informed consent form which was obtained from parents of all the children and healthy controls the individual participant data wouldn't be shared.